CLINICAL TRIAL: NCT00581750
Title: Molecular Genetic Basis of Invasive Breast Cancer Risk Associated With Lobular Carcinoma in Situ
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 01-135
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: Breast Cancer; Lobular Carcinoma; Invasive Breast Cancer
Keywords: Biopsy; Breast; 01-135
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Lobular | interventions — Histocompatibility Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Tissue
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- LCIS diagnosis: Patient with LCIS diagnosis
  Interventions: Other: Tissue specimen

INTERVENTIONS:
Other: Tissue specimen — Human tissues taken after the clinically indicated removal of these tissues from patients as part of their routine care.

SUMMARY:
This study is being done in order to better understand the biology of an abnormal lesion found in breast tissue called "lobular carcinoma in situ" (LCIS). We are interested in studying LCIS. The LCIS is not a cancer itself, but is a marker for an increased risk of cancer. We would like to look for LCIS in breast tissue removed during surgery from patients with cancer or at high risk for cancer. If LCIS is found, we will search for genes that are expressed (turned on or off) differently than in normal breast tissue. The identification of such genes would help us better understand the biology of LCIS, and its possible relationship to breast cancer.

DETAILED DESCRIPTION:
LCIS) is a monoclonal pathologic entity which is subject to characterization at the molecular genetic level, and that these molecular genetic alterations may be used to predict the subsequent development of invasive breast cancer. Prophylactic mastectomy specimens from women with multifocal LCIS, and invasive breast cancer specimens which display coexisting LCIS, will be examined for X-chromosome inactivation patterns and loss of heterozygosity to assess for monoclonality. If clonality is present, we will assess for microsatellite instability, and a microarray-based comparative genomic hybridization (CGH) technique will be used to identify genetic alterations present in LCIS. Lastly, LCIS biopsy specimens from untreated patients who, after follow-up did or did not develop invasive breast cancer, will be evaluated to determine whether the nature or extent of any identified genetic alterations can be correlated with the subsequent development of invasive breast cancer. We hypothesize that a fraction of LCIS lesions will reflect a monoclonal origin, that those lesions of monoclonal origin will display evidence of specific molecular genetic alterations, and that these specific alterations will correlate with the likelihood of the subsequent development of invasive breast carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* multifocal lobular carcinoma in situ treated with prophylactic mastectomy or lumpectomy
* invasive breast cancer (lobular or ductal) with coexisting lobular carcinoma in situ treated with mastectomy or lumpectomy
* biopsy proven, untreated lobular carcinoma in situ
* invasive lobular cancer with or without coexisting lobular carcinoma in situ treated with mastectomy or lumpectomy

Exclusion Criteria:

* no paraffin blocks available
* no residual lobular carcinoma in situ in paraffin blocks

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women seen at MSKCC breast clinic
Sampling Method: Non-Probability Sample
Enrollment: 550 (Estimated)
Dates: Start 2001-10; Primary Completion 2021-06-28 (Actual); Study Completion 2021-06-28 (Actual)

PRIMARY OUTCOMES:
To perform analyses using microarray-based gene expression profiling to determine whether a unique mRNA and microRNA gene expression profile distinguishes LCIS from normal breast epithelium and from invasive carcinoma. | 2 years

SECONDARY OUTCOMES:
To perform analyses using microarray-based mRNA and microRNA gene expression profiling to identify distinct molecular subtypes within LCIS. | 2 years
Deter the nature or extent of molecular genetic alterations in LCIS as asses by mRNA & microRNA microarray canbe correl with the risk of subsequent invas breast cancer in pts with class type LCIS & those with newly described histologic variants of LCIS. | 2 years
To prospectively follow patients diagnosed with newly described histologic variants of lobular carcinoma in situ, who do or do not undergo surgery for treatment or prevention, to better characterize this lesion and its behavior. | 2 years
To further characterize the invasive lobular breast cancers that develop in association with LCIS as assessed by standard histopathology and immunohistochemistry. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Pilewskie, M.D., Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center website — http://www.mskcc.org